CLINICAL TRIAL: NCT00278343
Title: A Phase 2 Study of AZD2171 in Recurrent or Persistent Ovarian, Peritoneal, or Fallopian Tube Cancer
Brief Title: Cediranib Maleate in Treating Patients With Persistent, Recurrent, or Refractory Advanced Ovarian Epithelial, Peritoneal Cavity, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03027; NCI-2012-03027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7129; PMH-PHL-037; PHL-037 (Other: Princess Margaret Hospital Phase 2 Consortium); 7129 (Other: CTEP); N01CM62209 (NIH); N01CM62201 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive cediranib maleate PO QD every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — 30mg given PO, daily
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well cediranib maleate works in treating patients with persistent, recurrent, or refractory advanced ovarian epithelial, peritoneal cavity, or fallopian tube cancer. Cediranib maleate may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Objective tumor response rate (complete plus partial response plus stable disease > 16 weeks as defined by the Response Evaluation Criteria in Solid Tumors [RECIST] criteria) in women with recurrent or refractory advanced ovarian or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. Time to disease progression, median survival time, and duration of overall cancer antigen (CA)-125 response.

OUTLINE:

Patients receive cediranib maleate orally (PO) once daily (QD) every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that has recurred or is refractory to initial therapy; patients must have received platinum-based chemotherapy before entry into this protocol
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan OR patients must have evidence of progression based on an elevated CA-125 (defined as a value of > 2 x upper limit of normal [ULN] documented on two separate determinations made > 2 weeks apart) if the physical exam is normal and CT scan of the chest/abdomen/pelvis, has a disease volume < 1 cm in maximum diameter
* Patients may have received no more than one prior chemotherapy regimen (i.e. initial first-line chemotherapy only)
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with borderline tumors or tumors of low malignant potential
* Patients with current bowel obstruction
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 30 days
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171 (cediranib maleate)
* Mean corrected QT (QTc) > 470 msec (with Bazett's correction) in screening electrocardiogram or history of familial long QT syndrome
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study, breastfeeding should be discontinued if the mother is treated with AZD2171
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Any significant abnormality noted in the electrocardiogram (ECG) within 14 days of treatment
* A New York Heart Association classification of III or IV (NOTE: patients classified as class II controlled with treatment may continue with increase monitoring)
* Conditions requiring concurrent use of drugs or biologics with proarrythmic potential; these drugs are prohibited during studies with AZD2171

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Hirte, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (28):
- United States (21):
  - City of Hope, Duarte, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - City of Hope Medical Group Inc, Pasadena, California
  - University of California at Davis Cancer Center, Sacramento, California
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Evanston Hospital CCOP, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Peoria Gynecologic Oncology, Peoria, Illinois
  - Oncology/Hematology Associates, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre-South Street, London, Ontario
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Cancer Centre (Ottawa Health Research Institute) Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec

REFERENCES:
- [Derived] Hirte H, Lheureux S, Fleming GF, Sugimoto A, Morgan R, Biagi J, Wang L, McGill S, Ivy SP, Oza AM. A phase 2 study of cediranib in recurrent or persistent ovarian, peritoneal or fallopian tube cancer: a trial of the Princess Margaret, Chicago and California Phase II Consortia. Gynecol Oncol. 2015 Jul;138(1):55-61. doi: 10.1016/j.ygyno.2015.04.009. Epub 2015 Apr 17. PMID 25895616

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cediranib Maleate): Patients receive cediranib maleate PO QD every 4 weeks in the absence of disease progression or unacceptable toxicity.
  cediranib maleate: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Platinum sensitive: 39 Platinum resistant: 35 Total # treated: 74
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 52
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Response Benefit (Complete Response or Partial Response or Stable Disease) Based on the RECIST/Rustin Criteria
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response(OR) = CR+PR
Time Frame: After 16 weeks
Population: Total # of Patients 74 PL-S (platinum sensitive) 39 patients PL-R (platinum resistant) 35 patients Confirmed PR PL-S group 9/39 patients Confirmed PR PL-R group 0/35 patients
Measure: Number; unit: participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 74
participants
  Platinum sensitive participants: number analyzed (Participants) | 39
  Platinum sensitive participants | 9
  Platinum resistant participants: number analyzed (Participants) | 35
  Platinum resistant participants | 0

2. Secondary Outcome: Time to Disease Progression
Description: Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: Up to 4 years
Population: Platinum sensitive cohort
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 47
months
  Platinum Sensitive Participants: number analyzed (Participants) | 23
  Platinum Sensitive Participants | 7.2 [3.9 to 9.4]
  Platinum Resistant Participants: number analyzed (Participants) | 25
  Platinum Resistant Participants | 3.7 [3.4 to 4.5]

3. Secondary Outcome: Overall Survival (OS) (Discontinued as of 4/25/2014)
Description: The Kaplan-Meier method will be used to estimate OS. Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: From date of radomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 32 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 74
months | 18.9 [13.5 to 31.5]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate PFS. Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions.
Time Frame: Time from start of treatment to time of progression, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 74
months | 4.9 [3.9 to 7]

5. Secondary Outcome: Duration of Overall CA-125 Response
Description: Confirmed response on CA125 - defined as reduction in level of pre-treatment sample by > 50%.
Time Frame: Up to 4 years
Population: 1 confirmed PR observed in PS group. Response will be defined as reduction in level of pre-treatment sample by > 50%.
  0 confirmed PR observed in PR group.
Measure: Number; unit: weeks
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 1
weeks
  Platinum sensitive participants | 108
  Platinum resistant participants: number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Toxicity Graded According to National Cancer Institution Common Terminology Criteria for Adverse Events Version 3.0
Time Frame: Up to 4 years
Population: Data were not collected.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 5/74
Other Adverse Events (participants affected / at risk) | 47/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=74)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=74)
Myocardial infarction (Cardiac disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 18 (18)
fatigue (General disorders) | 13 (13)
diarrhea (Gastrointestinal disorders) | 7 (7)
headache (Nervous system disorders) | 47 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less